CLINICAL TRIAL: NCT01042132
Title: Pathophysiological Effects of- and Inflammatory Response to Intramedullary Femoral Nailing in Patients With Femoral Shaft Fracture
Brief Title: Intramedullary Femoral Reaming, Human Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Principal Investigator, Elisabeth Ellingsen Husebye, MD, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02066
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2002-04

CONDITIONS: Pulmonary Complications; Organ Failure; Systemic Inflammatory Response Syndrome
Keywords: intramedullary reaming; inflammatory response; human; femoral shaft fracture; Reamer-irrigator-aspirator
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1) IMN and EF/IMN (Active Comparator): Two parts of the study are randomized;
  1)initial intramedullary reaming and primary external fixation with secondary intramedullary nailing
  Interventions: Procedure: the effect of delayed intramedullary reaming
- 2) TR and RIA (Active Comparator): Two parts of the study are randomized; 2)traditional reaming (TR)is compared to a new reaming device, RIA, which is a reamer connected to suction and flushing for prevention of increased intramedullary pressure
  Interventions: Procedure: the reaming of the femoral canal is performed with two different reaming devices

INTERVENTIONS:
Procedure: the effect of delayed intramedullary reaming — in one group intramedullary reaming and nailing is performed immediately, femoral fractures in the second group are external fixated and than secondary nailed.
  Arms: 1) IMN and EF/IMN
Procedure: the reaming of the femoral canal is performed with two different reaming devices — the reaming of the femoral canal is performed with two different reaming devices; a traditional reamer (TR)and the reamer-irrigator-aspirator (RIA)
  Arms: 2) TR and RIA

SUMMARY:
To what extent the cardiopulmonary and inflammatory response is affected by initial femoral intramedullary nailing in the already traumatized and inflammatory activated patient was analyzed in the present study with the attention to survey the additional burden of this operative treatment. The patients are monitored with a pulmonary catheter, and blood samples for coagulation, fibrinolysis, complement and cytokine response are withdrawn pre-, per- and postoperatively. The study is partly randomized 1)where delayed intramedullary nailing is compared with primary nailing of the femur, and 2) a new reaming technique (RIA) is compared with a standard reaming technique (TR).

DETAILED DESCRIPTION:
To what extent the cardiopulmonary and inflammatory response is affected by initial femoral intramedullary nailing in the already traumatized and inflammatory activated patient was analyzed in the present study with the attention to survey the additional burden of this operative treatment. The patients are monitored with a pulmonary catheter, and blood samples for coagulation, fibrinolysis, complement and cytokine response are withdrawn pre-, per- and postoperatively. The study is partly randomized 1)where delayed intramedullary nailing is compared with primary nailing of the femur, and 2) a new reaming technique (RIA) is compared with a standard reaming technique (TR).

ELIGIBILITY:
Inclusion Criteria:

* femoral shaft fracture suitable for intramedullary nailing
* < 24 hours postinjury

Exclusion Criteria:

* previous fracture of the femur
* pathological fracture
* femur deformities
* pregnancy
* previous intramedullary nailing or external fixation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-05; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
cardiopulmonary alterations | the first three postoperative days
coagulation, fibrinolytic and cytokine response | pre-, per- and first 3 days postoperatively

SECONDARY OUTCOMES:
fracture healing | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Olav Røise, MD, Study Director — Orthopedic Centre, Ullevaal University Hospital, Oslo, Norway
Locations (1):
- Orthopedic Center, Ullevål University Hopspital, Oslo, Norway